CLINICAL TRIAL: NCT06631027
Title: The Relationship Between Adherence to Mediterranean, DASH and MIND Diets and Cognitive Function in Older Adults
Brief Title: Dietary Adherence and Cognitive Function in Older Adults
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assit. of Prof, Ankara Yildirim Beyazıt University
Other Study IDs: AYBUELİBOL001
Record Dates: First submitted 2024-09-27; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Function; Mediterranean Diet; Dietary Approaches to Stop Hypertension; Elderly Population
Keywords: Cognitive Function; Mediterranean Diet; Elderly Health; DASH Diet; MIND Diet

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elderly Participants (65 years and older): This study focuses on a cohort of 1,027 elderly participants aged 65 years and older. The participants were assessed for their adherence to the Mediterranean, DASH, and MIND diets through a demographic questionnaire and dietary adherence scales. Cognitive function was evaluated using the Standardized Mini-Mental Test (SMMT). The study aims to explore the relationship between dietary patterns and cognitive health in this population.

SUMMARY:
This study aimed to evaluate the relationship between adherence to the Mediterranean, DASH, and MIND diets and cognitive function in elderly individuals. Data were collected from 1,027 participants aged 65 and older, using dietary assessment tools and the Standardized Mini Mental Test (SMMT), and were analyzed with SPSS 26.

DETAILED DESCRIPTION:
A total of 1027 elderly individuals aged 65 years and over were included in the study. Demographic questionnaire and Mediterranean diet adherence scale were administered to the individuals. Adherence to the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet was scored and food consumption was recorded for adherence to the Dietary Approaches to Stop Hypertension (DASH) diet. Standardised mini mental test (SMMT) was used to assess mental status. Data were analysed with SPSS 26 software.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 65 years and older.

Exclusion Criteria:

1. Individuals diagnosed with psychiatric or neurological diseases (e.g., dementia, Alzheimer's disease).

3. Individuals with alcohol or drug addiction. 4. Illiterate individuals.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community sample in Ankara, Turkey
Sampling Method: Non-Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Function Assessment | Basaline
  The primary outcome measure is the cognitive function of elderly individuals assessed using the Standardized Mini-Mental Test. The total Standardized Mini-Mental Test score is analyzed to evaluate the relationship between dietary adherence and cognitive function.The test is scored according to the answers given to each question and evaluated over 30 points in total. On a 30-point scale, a score of 24 and above indicates normal cognition, while a score below 24 indicates impaired cognitive function.

SECONDARY OUTCOMES:
Sociodemographic characteristics | basaline
  number and percentage
Mediterranean Diet Adherence Scale | Basaline
  Adherence to the Mediterranean Diet will be assessed using the Mediterranean Diet Adherence Scale. Scores will range from 0 to 14, with scores below 7 indicating non-compliance, 7-8 indicating acceptable compliance, and 9 and above indicating strict adherence to the Mediterranean diet.
Compliance with the Dietary Approaches to Stop Hypertension diet | Basaline
  Compliance with the Dietary Approaches to Stop Hypertension diet will be assessed using a 24-hour recall method to evaluate dietary intake. Scores range from 0 to 9, with scores of 4.5 or above indicating compliance with the DASH diet. This assessment will be used to explore the relationship between DASH diet adherence and cognitive function in elderly individuals.
Compliance with the Mediterranean-DASH Intervention for Neurodegenerative Delay diet | Basaline
  Compliance with the Mediterranean-DASH Intervention for Neurodegenerative Delay diet will be assessed by evaluating the frequency and portion sizes of key dietary components, Higher scores indicate greater adherence to the MIND diet. In this study, a median score of 7.5 will be used to categorize participants into two groups: those with a low level of adherence (score ≤7.5) and those with a high level of adherence (score >7.5).
Body Mass Index (BMI) | Basaline
  Kilograms per square meter (kg/m2)
Body weight | Basaline
  Body weight in kg
Height | Basaline
  Height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No